CLINICAL TRIAL: NCT01028547
Title: Antiemetic Efficacy and Safety of Dexamethasone in Patients Undergoing Caesarean Sections at Mulago Hospital
Brief Title: Antiemetic Efficacy and Safety of Dexamethasone in Obstetric Surgical Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Makerere University (Other)
Responsible Party: Dr Arthur Kwizera, Department of anaesthesia Makerere University College of health sciences
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PONVDEX
Record Dates: First submitted 2009-12-07; First posted 2009-12-09 (Estimated); Last update posted 2010-03-26 (Estimated); Status verified 2010-03

CONDITIONS: Postoperative Nausea and Vomiting
Keywords: PONV
MeSH Terms: conditions — Postoperative Nausea and Vomiting | interventions — Dexamethasone; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- dexamethasone 8mg (Active Comparator)
  Interventions: Drug: dexamethasone
- normal saline (Placebo Comparator)
  Interventions: Other: normal saline

INTERVENTIONS:
Drug: dexamethasone — single Bolus dose of dexamethasone 8mg
  Arms: dexamethasone 8mg
Other: normal saline — 2 ml 0.9% saline
  Arms: normal saline

SUMMARY:
This is a randomised controlled double blinded clinical trial to determine the antiemetic efficacy and safety of either 8 mg of dexamethasone or normal saline (placebo) given 1 hour before induction of either spinal or general anaesthesia in 2 arms (of 150 each).

ELIGIBILITY:
Inclusion Criteria:

* all woman above 18 years old presenting for obstetric surgery and have consented to study.

Exclusion Criteria:

* refusal/unable to consent,
* younger than 18 years old,
* hypertensive,
* diabetic,
* preeclamptic,
* sepsis,
* ASAIIIE plus.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 250 (Actual)
Dates: Start 2010-01; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
presence of post nausea and or vomiting | 24 hours

SECONDARY OUTCOMES:
perianal itching | 24 hours
hyperglycemia | 24 hours
hypertension | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Tindimwebwa J V B, MD, Study Director — Makerere university dept of anesthesia
Locations (1):
- Mulago National Refferal Hospital, Kampala, Uganda

REFERENCES:
- [Derived] Griffiths JD, Gyte GM, Popham PA, Williams K, Paranjothy S, Broughton HK, Brown HC, Thomas J. Interventions for preventing nausea and vomiting in women undergoing regional anaesthesia for caesarean section. Cochrane Database Syst Rev. 2021 May 18;5(5):CD007579. doi: 10.1002/14651858.CD007579.pub3. PMID 34002866